CLINICAL TRIAL: NCT01270347
Title: Phase 3, Open-label, Randomized Trial to Evaluate the Safety and Efficacy of MP-376 Inhalation Solution (Aeroquin) vs. Tobramycin Inhalation Solution (TIS) in Stable CF Patients
Brief Title: Trial of Aeroquin Versus Tobramycin Inhalation Solution (TIS) in Cystic Fibrosis (CF) Patients
Acronym: TIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mpex-209; 2010-019634-26 (EudraCT Number)
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Results first posted 2024-05-21 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aeroquin (Experimental): Aeroquin, Inhaled Levofloxacin (MP-376)
  Interventions: Drug: MP-376 (Levofloxacin Solution for Inhalation)
- TIS (Active Comparator): Tobramycin Inhalation solution (TIS) [TOBI® Novartis Pharmaceuticals]
  Interventions: Drug: TIS (Tobramycin Inhalation Solution)

INTERVENTIONS:
Drug: MP-376 (Levofloxacin Solution for Inhalation) — MP-376 (Aeroquin, Levofloxacin solution for Inhalation) 240 mg administered BID for 28-days treatment followed by 28 days off treatment
  Other Names: (Aeroquin, Levofloxacin solution for Inhalation)
  Arms: Aeroquin
Drug: TIS (Tobramycin Inhalation Solution) — Tobramycin Inhalation Solution administered BID over 3 consecutive cycles of 28-days treatment followed by 28 days off treatment
  Other Names: TOBI
  Arms: TIS

SUMMARY:
Patients with cystic fibrosis (CF) suffer from chronic infections of the lower respiratory tract that can be caused by one or multiple bacteria, including Pseudomonas aeruginosa, which has been particularly problematic to eradicate and been implicated as the major cause of morbidity and mortality in CF patients. Aerosol delivery of antibiotics directly to the lung increases the local concentrations of antibiotic at the site of infection resulting in improved antimicrobial effects compared to systemic administration. Bacterial resistance to current aerosol antibiotic treatments indicate a need for improved therapies to treat CF patients with pulmonary infections caused by multi-drug resistant Pseudomonas aeruginosa and other bacteria. High concentrations of MP-376 delivered directly to the lung are projected to have antimicrobial effects on even the most resistant organisms.

DETAILED DESCRIPTION:
This study will assess the comparative safety of MP-376 (Aeroquin) and Tobramycin Inhalation solution (TIS) [TOBI® Novartis Pharmaceuticals] over three consecutive cycles of 28-days treatment followed by 28-days off in stable CF patients with chronic P. aeruginosa lung infection. Efficacy data for MP-376 and TIS at the end of the first 28-day treatment period will also be compared, as well as explored over multiple treatment cycles.

Study patients participating in Mpex 209 will be given the option to participate in a six-month open label extension phase of the Mpex 209 protocol. The open label extension will allow enrolled patients to receive three additional courses of MP-376 (levofloxacin inhalation solution, Aeroquin™).

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria (selected):

* > 12 years of age
* Confirmed Diagnosis of Cystic Fibrosis
* Positive sputum culture for P. aeruginosa within the past 12 months
* Patients are able to elicit an FEV1 >/= 25% but </= 85% of predicted value at screening
* Have received at least 3 courses of inhaled tobramycin over the preceding 12 months
* Clinically stable with no changes in health status within the last 28 days
* Able to reproducibly produce sputum and perform spirometry

Exclusion Criteria (selected):

* Use of any nebulized or systemic antibiotics within 28 days prior to baseline
* History of hypersensitivity to fluoroquinolones or inhaled or systemic aminoglycosides including tobramycin or any excipients
* Evidence of acute upper within 10 days or lower respiratory infections within 28 days prior to dosing
* CrCl < 20 at Screening
* History of lung transplantation

Extension Portion of the Study: Patients enrolled in Mpex 209 are permitted to participate in the open label extension as long as they complete Visit 7 (Day 168), provide informed consent for participation in the open label extension of in the study and are clinically stable, as assessed by the Investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (123):
- United States (92):
  - Mobile, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Long Beach, California
  - Childrens Hospital, Los Angeles, California
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Denver, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Wilmington, Delaware
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Glenview, Illinois
  - Niles, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Manchester, New Hampshire
  - Livingston, New Jersey
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Albany Medical College #2, Albany, New York
  - Albany, New York
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma CF Center, Oklahoma City, Oklahoma
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Colchester, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Portsmouth, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- France (6):
  - Hôpital Pellegrin Enfants - CHU Bordeaux, Bordeaux
  - CRCM adultes et enfants Service des maladies respiratoires et pédiatrie 1 CHU- Arnaud de Villeneuve, Montpellier
  - Hôpital Cochin, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Haut-Lévêque CHU de Bordeaux, Pessac
  - CRCM adulte Hôpital Larrey-CHU de Toulouse, Toulouse
- Germany (11):
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitätskinderklinik Dresden Mukoviszidose-Ambulanz, Dresden
  - Universitätsklinikum Essen, Essen
  - Katharina-Kasper Kliniken GmbH St. Elisabethen-Krankenhaus Medizinische Klinik, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinik Gießen und Marburg GmbH Zentrum für Kinderheilkunde und Jugendmedizin, Gieben
  - Kinderärztliche Gemeinschaftspraxis Dr. H. E. Heuer, Dr. C. Runge, W. Sextro, Hamburg
  - Universitätsklinikum Kiel, Kiel
  - Dr. von Haunersches Kinderspital der Universität München Christiane Herzog Ambulanz, Munich
  - Ludwig-Maximilians Universität Klinikum Innenstadt, München
  - Universitätsklinik für Kinder- und Jugendmedizin, Tübingen
- Ireland (4):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - National Children's Hospital Tallaght, Dublin
  - St. Vincent's University Hospital, Dublin
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center Mount Scopus, Jerusalem
  - Schneider Childrens Medical Center of Israel, Petah Tikva
  - Safra Childrens Hospital, Sheba Medical Center, Ramat Gan
- United Kingdom (6):
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Castle Hill Hospital, Cottingham
  - St James's University Hospital, Leeds
  - King's College Hospital, London
  - University Hospital Llandough, Penarth, Penarth

REFERENCES:
- [Derived] Elborn JS, Flume PA, Cohen F, Loutit J, VanDevanter DR. Safety and efficacy of prolonged levofloxacin inhalation solution (APT-1026) treatment for cystic fibrosis and chronic Pseudomonas aeruginosa airway infection. J Cyst Fibros. 2016 Sep;15(5):634-40. doi: 10.1016/j.jcf.2016.01.005. Epub 2016 Feb 28. PMID 26935334

RESULTS

PARTICIPANT FLOW:
Groups:
- Tobramycin Inhalation Solution 300 mg/Aeroquin 240 mg: Participants received 300 mg of Tobramycin by inhalation route, BID over 3 consecutive 56-day cycles (28 days on treatment and 28 days off treatment) during core phase. Participants received 240 mg of Aeroquin by inhalation route, BID over 3 consecutive 56-day cycles (28days on treatment and 28 days off treatment) during extension phase.
- Aeroquin 240 mg/Aeroquin 240 mg: Participants received 240 milligrams (mg) of Levofloxacin by inhalation route, twice daily (BID) over 3 consecutive 56-day cycles (28 days on treatment and 28 days off treatment) during core phase. Participants received 240 mg of Aeroquin by inhalation route, BID over 3 consecutive 56-day cycles (28days on treatment and 28 days off treatment) during extension phase.
Period: Core Phase
Arm/Group | Tobramycin Inhalation Solution 300 mg/Aeroquin 240 mg | Aeroquin 240 mg/Aeroquin 240 mg
Started | 93 | 189
Completed | 83 | 166
Not Completed | 10 | 23
Not completed — Adverse Event | 1 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Miscellaneous | 8 | 14
Period: Extension Phase
Arm/Group | Tobramycin Inhalation Solution 300 mg/Aeroquin 240 mg | Aeroquin 240 mg/Aeroquin 240 mg
Started | 32 (Participants from US and Europe who completed core phase were allowed to enter into extension phase) | 56 (Participants from US and Europe who completed core phase were allowed to enter into extension phase)
Completed | 26 | 47
Not Completed | 6 | 9
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Miscellaneous | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants randomized in the study who received at least 1 dose of Levofloxacin inhalation solution or TIS.
Groups:
- Tobramycin Inhalation Solution 300 mg: Participants received 300 mg of Tobramycin by inhalation route, BID over 3 consecutive 56-day cycles (28 days on treatment and 28 days off treatment).
- Levofloxacin Inhalation Solution 240 mg: Participants received 240 mg of Levofloxacin by inhalation route, BID over 3 consecutive 56-day cycles (28 days on treatment and 28 days off treatment).
- Total: Total of all reporting groups
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg | Total
Number analyzed (Participants) | 90 | 182 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (11.05) | 28.3 (9.00) | 28.5 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 81 | 118
  Male | 53 | 101 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 14 | 17
  Not Hispanic or Latino | 87 | 168 | 255
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 87 | 174 | 261
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any unfavorable or unintended sign, symptom, or disease temporally associated with the use of a Study Drug, whether or not considered related to the Study Drug.
  An AE could potentially be a new disease, any untoward event, or an exacerbation of a pre-existing condition. AEs included, but were not limited to:
  Any symptom not previously reported by the patient (medical history) An exacerbation of a pre-existing illness An increase in frequency or intensity of a pre-existing episodic event or condition A condition first detected or diagnosed after Study Drug administration even though the condition may have been present before the start of the study Overdose of Study Drug
Time Frame: From start of study until end of the study (up to 168 days)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 90 | 182
participants | 90 | 180

2. Primary Outcome: Relative Change From Baseline in Percent Predicted Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 was the volume of air exhaled in first second of a forced expiration as measured by spirometer. Least squares (LS) mean and standard error (SE) were determined from an analysis of covariance model with terms for treatment, region (US, non-US), and age (12 to 18 years, > 18 years), and Baseline FEV1 (< 55%, . 55%).
Time Frame: Baseline, day 28
Population: Intent-to-treat population included all participants randomized in the study.
Measure: Least Squares Mean (Standard Error); unit: percent predicted FEV1
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 93 | 189
percent predicted FEV1 | 0.38 (1.262) | 2.24 (1.019)
Statistical Analysis 1: Comparison: Tobramycin Inhalation Solution 300 mg vs Levofloxacin Inhalation Solution 240 mg; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the LS mean difference 95% CI for relative change from Baseline to Day 28 in FEV1 percent predicted was > -4%; p = 0.1481, ANCOVA; LSMean difference = 1.86, 95% CI 2-sided [-0.66 to 4.39] — Estimates were determined from an analysis of covariance model with terms for treatment, region (US, non-US), and age (12 to 18 years, > 18 years), and Baseline FEV1 (< 55%, . 55%)

3. Secondary Outcome: Percent Change From Baseline in Average Expired Flow Over the Middle Half of The FVC Maneuver (FEF25-75)
Description: LSMean and SE were determined from an ANCOVA model with terms for treatment, region (US, non-US), age (12-18 years, >18 years), baseline FEV1 (<55%, >=55%), and baseline as a covariate.
Time Frame: Baseline, day 28
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 93 | 189
Percent change | 4.705 (8.8115) | 9.673 (2.2691)
Statistical Analysis 1: Comparison: Tobramycin Inhalation Solution 300 mg vs Levofloxacin Inhalation Solution 240 mg; Test type: Non-Inferiority — Non-inferiority is demonstrated if the lower limit of the LS mean difference 95% CI for relative change from baseline to Day 28 in FEV1 percent predicted is > -4%; p = 0.0830, ANCOVA; LSMean difference = 4.968, 95% CI 2-sided [-0.653 to 10.590] — Estimates are determined from an ANCOVA model with terms for treatment, region (US, non-US), age (12-18 years, >18 years), baseline FEV1 (<55%, >=55%), & baseline as a covariate

4. Secondary Outcome: Percent Change From Baseline in Forced Vital Capacity (FVC)
Description: as for outcome 3
Time Frame: Baseline, day 28
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 93 | 189
Percent change | -1.152 (0.9191) | 0.417 (0.7441)
Statistical Analysis 1: Comparison: Tobramycin Inhalation Solution 300 mg vs Levofloxacin Inhalation Solution 240 mg; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.0945, ANCOVA; LSMean difference = 1.570, 95% CI 2-sided [-0.272 to 3.411] — Estimates are determined from a repeated measures model with terms for treatment, visit, the interaction between treatment group and visit, region (US, non-US), age (12-18 years, >18 years), baseline FEV1 (<55%, >=55%), and baseline as a covariate

5. Secondary Outcome: Number of Participants in Each Category of Relative Change in Percent Predicted FEV1
Description: FEV1 was the volume of air exhaled in first second of a forced expiration as measured by spirometer.
Time Frame: Day 28
Population: ITT population with available data at specified timepoint.
Measure: Number; unit: participants
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 88 | 172
participants
  Moderate decline (decline >=10%, death, or lung transplant) | 16 | 30
  Mild decline (0% < decline < 10%) | 26 | 59
  Mild improvement (0% <= improvement < 10%) | 37 | 72
  Moderate improvement (10% <= improvement < 20%) | 6 | 6
  Significant improvement (improvement >= 20%) | 3 | 5

6. Secondary Outcome: Number of Participants in Each Category of Percent Change From Baseline in FEV1
Description: FEV1 was the volume of air exhaled in first second of a forced expiration as measured by spirometer.
Time Frame: Day 28
Population: ITT population with available data.
Measure: Number; unit: participants
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 93 | 189
participants
  Moderate decline (decline >=10%, death, or lung transplant) | 13 | 9
  Mild decline (0% < decline < 10%) | 31 | 48
  Mild improvement (0% <= improvement < 10%) | 37 | 103
  Moderate improvement (10% <= improvement < 20%) | 8 | 26
  Significant improvement (improvement >= 20%) | 4 | 3

7. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa Sputum Density
Description: Pseudomonas aeruginosa density was measured as log10 colony-forming units [CFU] per gram sputum.
Time Frame: Baseline, day 28
Population: ITT population with available data at specified time point
Measure: Least Squares Mean (Standard Error); unit: log10 CFU per gram
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 79 | 161
log10 CFU per gram | -1.19 (0.243) | -0.75 (0.196)
Statistical Analysis 1: Comparison: Tobramycin Inhalation Solution 300 mg vs Levofloxacin Inhalation Solution 240 mg; Test type: Non-Inferiority — Non-inferiority is demonstrated if the lower limit of the LS mean difference 95% CI for relative change from baseline to Day 28 in Pseudomonas Aeruginosa Sputum Density is > -4%; p = 0.0530, ANCOVA; LSMean difference = 0.44, 95% CI 2-sided [-0.01 to 0.88] — Estimates are determined from an ANCOVA model with terms for treatment, region (US, non-US), age (12-18 years, >18 years), baseline FEV1 (<55%, >=55%), and baseline organism log density

8. Secondary Outcome: Number of Participants in Each Category of Change From Baseline in Pseudomonas Aeruginosa Sputum Density
Description: Pseudomonas aeruginosa density was measured as log10 colony-forming units [CFU] per gram sputum.
Time Frame: Baseline, day 28
Population: ITT population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 79 | 161
participants
  > 1.5 log decrease | 20 | 32
  >= 0.5 to <= 1.5 log decrease | 17 | 36
  < 0.5 decrease and < 0.5 log increase | 34 | 61
  >= 0.5 to <= 1.5 log increase | 4 | 18
  > 1.5 log increase | 4 | 14

9. Secondary Outcome: Change From Baseline in the Respiratory Domain of the Cystic Fibrosis Questionnaire Revised (CFQ-R)
Description: The Cystic Fibrosis Questionnaire (CFQ-R) is a disease-specific instrument that measures health-related quality of life (HRQOL) for adolescents and adults with cystic fibrosis (CF). Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, day 28
Population: ITT population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 91 | 186
Score on a scale | -1.31 (1.576) | 1.88 (1.278)
Statistical Analysis 1: Comparison: Tobramycin Inhalation Solution 300 mg vs Levofloxacin Inhalation Solution 240 mg; Test type: Non-Inferiority — Non-inferiority is demonstrated if the lower limit of the LS mean difference 95% CI for relative change from baseline to Day 28 in Respiratory Domain of the CFQ-R is > -4%; p = 0.0463, ANCOVA; LSMean difference = 3.19, 95% CI 2-sided [0.05 to 6.32] — Estimates are determined from an ANCOVA model with terms for treatment, region (US, non-US), age (12-18 years, >18 years), baseline FEV1 (<55%, >=55%), and baseline value

10. Secondary Outcome: Number of Participants in Each Category of Change From Baseline in the Respiratory Domain of CFQ-R
Description: as for outcome 9
Time Frame: Baseline, day 28
Population: ITT population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Tobramycin Inhalation Solution 300 mg | Levofloxacin Inhalation Solution 240 mg
Number analyzed (Participants) | 91 | 186
participants
  >= 4 increase | 25 | 81
  < 4 increase and < 4 decrease | 32 | 49
  >= 4 decrease | 34 | 56

ADVERSE EVENTS:
Time Frame: From start of study until end of the study (up to 168 days)
Description: Safety Population
Groups:
- Tobramycin Inhalation Solution 300 mg - Core Phase: Participants received 300 mg of Tobramycin by inhalation route, BID over 3 consecutive 56-day cycles (28 days on treatment and 28 days off treatment) during core phase.
- Aeroquin 240 mg - Core Phase: Participants received 240 mg of Levofloxacin by inhalation route, BID over 3 consecutive 56-day cycles (28 days on treatment and 28 days off treatment) during core phase.
- Aeroquin 240 mg - Extension Phase: Participants received 240 mg of Aeroquin by inhalation route route, BID over 3 consecutive 56-day cycles (28 days on treatment and 28 days off treatment) during extension phase.
Arm/Group | Tobramycin Inhalation Solution 300 mg - Core Phase | Aeroquin 240 mg - Core Phase | Aeroquin 240 mg - Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/182 | 0/88
Serious Adverse Events (participants affected / at risk) | 29/90 | 40/182 | 22/88
Other Adverse Events (participants affected / at risk) | 88/90 | 180/182 | 82/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tobramycin Inhalation Solution 300 mg - Core Phase (N=90) | Aeroquin 240 mg - Core Phase (N=182) | Aeroquin 240 mg - Extension Phase (N=88)
Disease progression (General disorders) | 24 (35) | 31 (39) | 16 (18)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (3) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Solution 300 mg - Core Phase (N=90) | Aeroquin 240 mg - Core Phase (N=182) | Aeroquin 240 mg - Extension Phase (N=88)
Abdominal pain (Gastrointestinal disorders) | 6 | 7 | 1
Nausea (Gastrointestinal disorders) | 7 | 11 | 3
Disease progression (General disorders) | 57 | 98 | 45
Exercise tolerance decreased (General disorders) | 14 | 23 | 11
Fatigue (General disorders) | 25 | 58 | 18
Malaise (General disorders) | 5 | 1 | 3
Pyrexia (General disorders) | 10 | 17 | 6
Nasopharyngitis (Infections and infestations) | 11 | 17 | 11
Sinusitis (Infections and infestations) | 8 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 1
Blood glucose increased (Investigations) | 7 | 4 | 0
Breath sounds abnormal (Investigations) | 1 | 1 | 5
Forced expiratory volume decreased (Investigations) | 15 | 17 | 14
Pulmonary function test decreased (Investigations) | 8 | 14 | 8
Weight decreased (Investigations) | 36 | 57 | 35
Decreased appetite (Metabolism and nutrition disorders) | 16 | 23 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 10 | 4
Dysgeusia (Nervous system disorders) | 0 | 46 | 12
Headache (Nervous system disorders) | 6 | 11 | 3
Sinus headache (Nervous system disorders) | 13 | 35 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 105 | 40
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 15 | 21 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 | 29 | 12
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 28 | 59 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 14 | 4
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 18 | 49 | 14
Rales (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 7
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 32 | 68 | 32
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 16 | 26 | 8
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 40 | 95 | 37
Rash (Skin and subcutaneous tissue disorders) | 7 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other